CLINICAL TRIAL: NCT02034747
Title: A Multicenter, Randomized, Comparison, Open-label, Phase IV Study to Assess the Efficacy and Safety of Advagraf® Switching From Cyclosporine Between the Group That Was Treated With a 50% Reduced Corticosteroid and the Group With Maintained Corticosteroid for Stable Kidney Transplant Recipients
Brief Title: A Study to Assess the Efficacy and Safety of Advagraf® Switching From Cyclosporine Between the Group That Was Treated With a 50% Reduced Corticosteroid and the Group With Maintained Corticosteroid for Stable Kidney Transplant Recipients
Acronym: COSMOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADV-KT-13-01
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplant
Keywords: Immunosuppressive regimen; Advagraf; kidney transplant; Corticosteroid
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corticosteroid with the 50% reduced dose (Experimental): oral
  Interventions: Drug: Advagraf; Drug: Corticosteroid
- Corticosteroid with the maintained dose (Active Comparator): oral
  Interventions: Drug: Advagraf; Drug: Corticosteroid

INTERVENTIONS:
Drug: Advagraf — oral
Drug: Corticosteroid — oral

SUMMARY:
This study is a multicenter, randomized, comparison, open-label, phase IV study in kidney transplant recipients whose immunosuppressive regimen is converted from Cyclosporine with corticosteroid to Advagraf® with corticosteroid. The eligible patients will be randomized into either Arm 1 or Arm 2. The Arm 1 will be reduced corticosteroid slowly until 50% lower dose from 4 weeks to 12 weeks in the Advagraf®-based immunosuppressive regimen, and the Arm 2 will receive the same corticosteroid dose for 24 weeks with Advagraf ®.

DETAILED DESCRIPTION:
The primary objective is to assess the changes in the GFR after 24 weeks of treatment between the group that was reduced corticosteroid slowly until 50% lower dose from 4 weeks to 12 weeks and the group with maintained corticosteroid in stable kidney transplant subjects whose regimen was converted from a CyA-based immunosuppressive regimen with corticosteroid to an Advagraf®-based immunosuppressive regimen with corticosteroid for kidney transplant subjects whose regimen was converted from a CyA-based immunosuppressive regimen.

The secondary objective is to assess the creatinine clearance rate, acute rejection, satisfaction of medication and safety of the group with a 50% reduced dose of corticosteroid and the group in which the Advagraf ®-based immunosuppressive regimen with maintained corticosteroid.

ELIGIBILITY:
Inclusion Criteria:

* Had a kidney transplant at least 12 months before his/her enrollment in this study (including a kidney retransplantation).
* Underwent a CyA-based immunosuppressive regimen since his/her last transplantation. The CyA dose remained unchanged during the last four weeks before the subject's enrollment.
* The immunosuppressive regimen (combination of medications) remained unchanged for a minimum of four weeks before the subject's enrollment.
* GFR≥30 mL/min

Exclusion Criteria:

* Had received an organ transplant other than a kidney
* Had an acute rejection episode within 12 weeks before his/her enrollment in this study, or had an acute rejection episode within 24 weeks before his/her enrollment in this study that required anti-lymphocyte antibody therapy
* Had been diagnosed with new-onset malignancy after his/her transplantation, except for basocellular or squamous cell carcinoma of the skin that had been treated successfully
* The subject received a kidney transplant from full-HLA identical donor
* Known to have FSGS or MPGN Type II as an underlying disease
* Has elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin levels ≥ 2 times the upper value of the normal range of the investigated site
* Has liver cirrhosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2015-11-07 (Actual); Study Completion 2015-11-07 (Actual)

PRIMARY OUTCOMES:
Change in the GFR before the treatment (baseline) to that on Week 24 | Baseline and Week 24

SECONDARY OUTCOMES:
Change in the GFR before the treatment (baseline) to that on Week 12 | Baseline and Week 12
Change in the creatinine clearance before the treatment (baseline) to those on Weeks 12 and 24 | Baseline, Week 12 and Week 24
Incidence of acute rejection | Up to Week 24
Safety assessed by the incidence of adverse events, vital signs and Lab-test | Up to Week 24
Physical examinations including cyclosporine related cosmetic side effect | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (9):
- South Korea (9):
  - Busan
  - Chungcheongnam-do
  - Daegu
  - Gyeonggi-do
  - Incheon
  - Jeollabuk-do
  - Jeollanam-do
  - Seoul
  - Ulsan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=197